CLINICAL TRIAL: NCT01063933
Title: A Pharmacokinetic/Pharmacodynamic and Safety Evaluation of Investigational Intravenous Peramivir in Children With Influenza Disease (CASG 117)
Brief Title: Pharmacokinetic/Pharmacodynamic and Safety Evaluation of Intravenous Peramivir in Children With Influenza
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Director ORA, HHS/NIAID/DMID
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-0064; BCX1812-205, CASG 117; N01AI30025C; N01AI30025 (NIH)
Record Dates: First submitted 2010-02-04; First posted 2010-02-05 (Estimated); Last update posted 2011-11-11 (Estimated); Status verified 2010-01

CONDITIONS: Influenza
Keywords: influenza, Peramivir, children, pharmacokinetic, pharmacodynamic
MeSH Terms: conditions — Influenza, Human | interventions — peramivir

ARMS (7):
- Cohort I (Experimental): Cohort I: >/= 12 years to < 18 years. Peramivir administered daily for five days or until the day of hospital discharge, whichever comes first.
  Interventions: Drug: Peramivir
- Cohort II (Experimental): Cohort II: >/= 6 years to < 12 years
  Interventions: Drug: Peramivir
- Cohort III (Experimental): Cohort III: >/= 2 years to < 6 years
  Interventions: Drug: Peramivir
- Cohort V (Experimental): Cohort V: >/= 91 days to < 181 days
  Interventions: Drug: Peramivir
- Cohort VII (Experimental): Cohort VII: birth to < 31 days
  Interventions: Drug: Peramivir
- Cohort VI (Experimental): Cohort VI: >/= 31 days to < 91 days
  Interventions: Drug: Peramivir
- Cohort IV (Experimental): Cohort IV: >/= 181 days to < 2 years
  Interventions: Drug: Peramivir

INTERVENTIONS:
Drug: Peramivir — Peramivir is a liquid for parenteral administration. Cohort I: Peramivir, 10 mg/kg intravenously (IV) every day (QD) (maximum of 600 mg/day) for 5 days or until hospital discharge, whichever comes first. Cohort II: Peramivir 12 mg/kg IV QD (maximum of 600 mg/day) for 5 days or until hospital discharge, whichever comes first. Cohort III: Peramivir 16 mg/kg QD (maximum of 600 mg/day) for 5 days or until hospital discharge, whichever comes first. Proposed doses for subjects in Cohorts IV, V, VI, and VII are 18, 18, 14 and 12 mg/kg, respectively, IV, QD for 5 days or until hospital discharge, whichever comes first. IV peramivir will be administered over 60 minutes.

SUMMARY:
The purposes of this study are to evaluate the pharmacokinetics (affect the body has on a drug), and pharmacodynamics (affect the drug has on the body) and safety of an experimental intravenous (within a vein) flu medication, peramivir, in children. Participants will include 63 hospitalized children with confirmed flu. Children will be grouped according to age and younger children will not receive drug until safety data from the groups of older children are reviewed. Hospitalized children may receive up to 5 doses of peramivir. Study procedures include: nasal/throat swabs, reporting any experienced side effects, physical examination including assessment of the nervous system, and blood sample collection. Participants will be involved in study related procedures for up to 28 days.

DETAILED DESCRIPTION:
Infants and young children are at greatest risk of mortality from epidemic influenza. Influenza medications currently approved for use in the United States are administered orally or via inhalation. Availability of a parenteral influenza medication could be of great importance in medical and public health responses to both seasonal and pandemic influenza. Peramivir is an experimental parenteral influenza drug that is in advanced stages of clinical development. The primary objective of this study is to define the pharmacokinetics (PK) of peramivir in children with confirmed influenza. The secondary objectives are to: assess the safety and tolerability of intravenous (IV) peramivir in children with influenza; assess viral dynamics as a function of drug PK; and assess virus susceptibility to peramivir. This study is a prospective, open-label, age-stratified PK/pharmacodynamic (PD) and safety evaluation of investigational IV peramivir in hospitalized children with influenza infection who are unable to receive or have failed at least three days oseltamivir or zanamivir therapy. A minimum of 63 children with confirmed influenza will be enrolled into 1 of 7 age cohorts: Cohort I (>= 12 years to < 18 years); Cohort II (>= 6 years to < 12 years); Cohort III (>= 2 years to < 6 years); Cohort IV (>= 181 days to < 2 years); Cohort V (>= 91 days to < 181 days); Cohort VI (>= 31 days to < 91 days) and Cohort VII (Birth to < 31 days). Only hospitalized children will be enrolled. At study onset, Cohorts I, II and III (children from >=2 years to < 18 years of age) will be enrolled initially. When PK and safety data from 9 total subjects enrolled Cohort I, Cohort II and/or Cohort IIII are available and reviewed by the study's Data and Safety Monitoring Board (DSMB), Cohorts IV-VII will be opened for enrollment. The initial doses selected for use were based on modeling and from a recently completed clinical trial study of a fixed dose (10 mg/kg) of peramivir in pediatric patients with influenza. In the current study, PK data will be obtained in a real time basis, and doses in each cohort may be modified if the target exposure [area under the curve (AUC) 24] falls outside of a pre-specified range. Additional enrollments may be allowed if the dose requires modification in a given cohort. In the event of a public health emergency, the National Institutes of Health (NIH), DSMB, or Food and Drug Administration (FDA) may that all cohorts be open for enrollment. Subjects will receive IV Peramivir once daily for 5 days or until the day of hospital discharge, whichever comes first, and PK blood draws will be obtained around the second dose. In addition to PK and PD, this study will carefully assess clinical disease course and adverse events (AEs), including neurologic AEs. Safety evaluations also will include neurologic assessments, general physical assessments, and AE and serious adverse event (SAE) reporting. Sequential nasopharyngeal specimens will be obtained for virologic assessments, including viral cultures, polymerase chain reaction (PCR) for viral ribonucleic acid (RNA) (quantitative), and analysis of antiviral resistance.

ELIGIBILITY:
Inclusion Criteria: -Signed informed consent from parent(s) or legal guardian(s), and signed informed assent as age appropriate. -Age: Cohort I:>/= 12 years to < 18 years. Cohort II: >/= 6 years to < 12 years. Cohort III: >/= 2 years to < 6 years. Cohort IV: >/= 181 days to < 2 years. Cohort V: >/= 91 days to < 181 days. Cohort VI: >/= 31 days to < 91 days. Cohort VII: Birth to < 31 days -Confirmed laboratory diagnosis of influenza by viral culture, polymerase chain reaction (PCR), or rapid influenza diagnostic test. -Hospitalized with influenza or complications of influenza -Subject cannot tolerate oral or inhaled influenza antiviral therapy, or has not responded to at least 3 days of oral or inhaled influenza antiviral therapy, as determined by the physician. -Females of childbearing potential must have one of the following: a. Subject has been sexually abstinent for the 4 weeks prior to date of screening evaluation and is willing to remain abstinent through 4 weeks after study drug administration b. Subject has been using oral contraceptives or other form of hormonal birth control for 3 months prior to the study and will continue to use through 4 weeks after study-drug discontinuation c. Subject has been using an intra-uterine device, or adequate double-barrier method (such as condom or diaphragm with spermicide) as birth control for 4 weeks prior to date of screening and will continue use through 4 weeks after study drug administration d. Subject is surgically sterile (e.g., hysterectomy, tubal ligation) -Sexually active males must ensure that their female partners of childbearing potential will utilize approved contraceptive methods to avoid pregnancy Exclusion Criteria: -Currently receiving peritoneal dialysis. -Currently requiring extracorporeal membrane oxygenation (ECMO). -Imminent demise. -Documented H275Y mutation (note: it is unlikely that resistance testing will have been completed for most subjects). -New onset seizure disorder with this acute illness. -Suspicion of significant renal impairment (e.g., polycystic renal disease, nephrectomy, renal transplantation within the past 6 months, renal agenesis, chronic renal failure, anuria). -Pregnancy (positive urine or serum pregnancy test at screening evaluation for females of childbearing potential). -Females who are breastfeeding. -Inability to comply with protocol-required procedures. -Presence of any pre-existing condition that, in the opinion of the investigator, would place the subject at an unreasonable increased risk through participation in this study. -Alternate explanation for clinical findings, as determined by the investigator.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Primary Completion 2011-08 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Peramivir dose that provides area under the curve (AUC)24 between 60 microgram (mcg) hour(hr)/liter (L) and 94 mcg hr/L. | Within 15 minutes prior to dosing, and at the following timepoints measured from the time of the start of the infusion: 1-1.25 hours (end of infusion), 2-3 hours, 5-7 hours, 10-12 hours, and 22-24 hours post-dosing.
Pharmacokinetic parameters for peramivir, including AUC24, maximum serum concentration (Cmax), half-life (T1/2), Clearance (CL), and time to maximum concentration (Tmax). | Within 15 minutes prior to dosing, and at the following timepoints measured from the time of the start of the infusion: 1-1.25 hours (end of infusion), 2-3 hours, 5-7 hours, 10-12 hours, and 22-24 hours post-dosing.

SECONDARY OUTCOMES:
Safety: overall incidence of adverse events. | Day 1 to Day 28
Safety: the incidence of grade 3-4 adverse events or severe adverse events. | Day 1 to Day 28
Safety: the incidence of adverse events considered to be related to study treatment. | Day 1 to Day 28
Safety: the incidence of adverse events leading to discontinuation of study drug. | Day 1 to Day 28
Virologic: proportion of subjects who are negative for viral ribonucleic acid (RNA) by reverse transcriptase-polymerase chain reaction (PCR). | Day 3, 5, and 10.
Virologic: incidence of treatment emergent peramivir resistant virus. | Study days 1, 3, 5, and 10.
Virologic: time to no detectable viral ribonucleic acid (RNA) by polymerase chain reaction (PCR). | Study days 1, 3, 5, and 10.
Virologic: quantitative viral load over time. | Study days 1, 3, 5, and 10.
Safety: the incidence of severe or grade 3 and 4 treatment related adverse events. | Day 1 to Day 28
Safety: the incidence of treatment-related serious adverse events. | Day 1 to Day 28
Safety: the incidence of serious adverse events and deaths. | Day 1 to Day 28

CONTACTS AND LOCATIONS:
Locations (29):
- United States (29):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Children's Hospital of Orange County, Orange, California
  - Stanford University, Stanford, California
  - The Children's Hospital - Denver, Colorado, Denver, Colorado
  - Childrens National Medical Center, Washington D.C., District of Columbia
  - University of South Florida, Tampa, Florida
  - University of Louisville, Louisville, Kentucky
  - Tulane University, New Orleans, Louisiana
  - Louisiana State University, Shreveport, Louisiana
  - Boston Medical Center, Boston, Massachusetts
  - University of Massachusetts, Worcester, Massachusetts
  - Washington University in St. Louis, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - The Children's Hospital at Saint Peter's University Hospital, New Brunswick, New Jersey
  - North Shore-Long Island Jewish Health System, Manhasset, New York
  - NYU School of Medicine, New York, New York
  - New York Presbyterian Hospital-Weill Medical College of Cornell University, New York, New York
  - University of Rochester, Rochester, New York
  - SUNY at Stony Brook, Stony Brook, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - MetroHealth Medical Center, Cleveland, Ohio
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Vanderbilt University, Nashville, Tennessee
  - The University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas